CLINICAL TRIAL: NCT04192864
Title: Comparison Between the Lingually Based and the Buccally Based Triangular Flap Design in the Surgical Removal of Impacted Mandibular Third Molars (Randomized Split Mouth Clinical Trial)
Brief Title: Comparison Between the Lingually Based and the Buccally Based Triangular Flap Design in the Surgical Removal of Impacted Mandibular Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Triagnular flap design
Record Dates: First submitted 2019-12-07; First posted 2019-12-10 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Tooth, Impacted
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: this study involved 20 patient with bilaterally mesially angulated impacted third molar (class II position B). One side was surgically removed using the lingually based triangular flap and the other side was surgically removed using the bucally based triangular flap
Who Masked: Participant
Masking Description: This study was a single blinded trial, where the participants did not know the technique used in each side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lingually based triangular flap (Experimental)
  Interventions: Procedure: Lingually based triangular flap
- Buccally based triangular flap (Active Comparator)
  Interventions: Procedure: Buccally based triangular flap

INTERVENTIONS:
Procedure: Lingually based triangular flap — A lingually based triangular flap was used to remove the impacted third molar. An incision was made adjacent to the distal surface of the mandibular second molar and extended along the sulcus to the distobuccal corner of the mandibular second molar, an oblique vestibular incision was made and extended into the vestibular fornix of the mandible. Aligned with the mesiobuccal cusp of the second molar.
  It was continued posterosuperior towards the anterior border of the mandibular ramus An incision will be made from the anterior border of the mandibular ramus to the distal surface of the mandibular second molar.
  Arms: Lingually based triangular flap
Procedure: Buccally based triangular flap — The impacted teeth was removed using a buccal based triangular flap. It will be extended along the sulcus to the distobuccal corner of the second molar . The incision was continuous, with a relieving vertical incision, oblique into the mandibular vestibular fornix, aligned with the mesiobuccal cusp of the second molar.
  Arms: Buccally based triangular flap

SUMMARY:
The primary objective of this study was to compare between the lingually based triangular flap with the buccally based triangular flap in the surgical removal of impacted mandibular third molars.

DETAILED DESCRIPTION:
Many flap designs used for impacted third molar surgery do not place the mucoperosteal incision on sound bone, as they involve incisions that are placed on the extraction socket resulting in higher incidence of mucosal dehiscence, followed by secondary wound healing

This study involved 20 patient with bilaterally mesially angulated impacted third molar (class II position B). One side was surgically removed using the lingually based triangular flap and the other side was surgically removed using the bucally based triangular flap

ELIGIBILITY:
Inclusion Criteria:

Presence of impacted third molar that is misally angulated and retained in bone (class II position B).

Exclusion Criteria:

* Patients with a history of systemic disease (diabetes, renal failure, immunocompromised patients, cardiac patients and patients taking radiotherapy or chemotherapy )
* Compromised dental and periodontal status
* Heavy Smoking.
* Pregnancy or lactation

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-10-13 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain using Visual Analogue Scale (VAS) | 7 days
  Pain was assessed through on a 10-point Visual Analogue Scale (VAS). (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Postoperative Edema | 7 days
  For the objective evaluation of swelling, five distances were measured
  * The distance from the mandibular angle to the lateral corner of the mouth
  * The distance from the mandibular angle to the nasal alar curvature
  * The distance from the mandibular angle to the lateral canthus of the eye
  * The distance from the tragus to the soft tissue pogonion
  * The distance from the tragus to the lateral corner f the mouth
Trismus Assessment | 7 days
  Trismus was assessed by measuring the maximum inter-incisional opening (in millimeters) the distance between the incisal edge of the upper and lower central incisor using caliber.
Wound healing/ Presence of alveolar osteitis | 21 days
  The presence of alveolar osteitis (dry socket) will be determined clinically using BLUM'S criteria. Wound healing was assessed and recorded depending on the absence or presence of dehiscence, every opening along the incision will be recorded as dehiscence , dental tweezers will be used to identify it.

CONTACTS AND LOCATIONS:
Overall Officials: Nesma M El-Atris, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Saeeda Osman, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Ahmed Swedan, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Garcia Garcia A, Gude Sampedro F, Gandara Rey J, Gallas Torreira M. Trismus and pain after removal of impacted lower third molars. J Oral Maxillofac Surg. 1997 Nov;55(11):1223-6. doi: 10.1016/s0278-2391(97)90172-5. PMID 9371111
- [Background] Conrad SM, Blakey GH, Shugars DA, Marciani RD, Phillips C, White RP Jr. Patients' perception of recovery after third molar surgery. J Oral Maxillofac Surg. 1999 Nov;57(11):1288-94; discussion 1295-6. doi: 10.1016/s0278-2391(99)90861-3. PMID 10555792
- [Background] Azaz B, Shteyer A, Piamenta M. Radiographic and clinical manifestations of the impacted mandibular third molar. Int J Oral Surg. 1976 Aug;5(4):153-60. doi: 10.1016/s0300-9785(76)80037-3. PMID 821867